CLINICAL TRIAL: NCT04290949
Title: Platelet Indices in Patients Undergoing Primary Percutaneous Coronary Intervention :Its Relation to the Severity of Coronary Artery Disease and Its Prognostic Value
Brief Title: Platelet Indices in Patients Undergoing Primary PCI and Its Prognostic Value
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ishraq Hosny Abd El-Hameed Hassan, Critical Care Unit, Internal Medicine Department, Assiut University
Other Study IDs: Platelet indices in acute MI
Record Dates: First submitted 2019-09-30; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the platelet indices in patients undergoing primary percutaneous coronary intervention and its relation to the severity of coronary artery disease and short term clinical outcomes

DETAILED DESCRIPTION:
Acute coronary syndromes (ACS) is a type of acute coronary artery disease (CAD), It is a highly prevalent group of emergency diseases, associated with high morbidity and mortality (1)

ACS include ST- elevation Myocardial Infarction (STEMI), non ST-Elevation Myocardial Infarction (NSTEMI) and Unstable Angina (UA) (2).

ACS characterized by plaque rupture and acute thrombosis formation in the coronary arteries (3)

platelet morphology and function have vital roles in the pathogenesis of many diseases related to coagulation, thrombosis, inflammation, and endothelial dysfunction (4)

Platelets play a crucial role in thrombotic episodes, its activation is acritical factor in the creation and evolution of atherothrombosis. (5)

Not only platelets are essential for the thrombotic vascular occlusion at the ruptured atherosclerotic plaque but also they contribute to the obstruction and impairment of coronary micro circulation (6).

Risk stratification plays a crucial role in the management of patients with ACS (7).

Patients estimated to be at higher risk may be managed with earlier and more aggressive treatment, whereas those with lower risk may be managed with less intensive treatment (8).

Many biomarkers have been evaluated, and various scores have been created for risk stratification of ACS patients (9)

Mean platelet volume (MPV) has been proposed as a primary marker for platelet activation, as larger sized platelets have been associated with higher pro-thrombotic risk, and its measurement is easy and time effective (10-14)

* So It may elevate in patients with ACS and its role, It could be a useful bio marker of risk of stratification (15)
* Platelet Distribution Width (PDW) measured on admission is a cheap and generally available biomarker which allows for predicting the development of heart failure in patients with ACS after PCI (16)

showed that an increased level of PDW was related to the severity of CAD in patients with ACS (17).

Numerous studies support the association of Mean platelet volume (MPV) with adverse cardiac outcomes as restenosis stent thrombosis in patients with ACS (19-24) al.2011

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) that presented with acute ST elevation myocardial infarction

Exclusion Criteria:

1. Cardiomyopathy,
2. Previous revascularization procedure
3. Any history of bleeding diathesis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients presented with acute myocardial infarction who undergoing primary percutaneous intervention
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
the severity of coronary artery disease and short term clinical outcomes | follow up patients 6 monthes
  Platelet indices as mean Platelet Volume (MPV)in femtoliter , platelet distribution width (PDW) (FL)% and (PCT)% May be larger and could be a risk of Stratification in patients undergoing primary percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El din Abd El Moniem, Professor, Study Director — Critical Care Unit, Internal Medicine Department

IPD SHARING:
Plan to Share IPD: Undecided